CLINICAL TRIAL: NCT00054002
Title: Surgery and Intracavitary Photodynamic Therapy (PDT) for the Treatment of Malignant Pleural Mesothelioma; The Use of Light Delivery Fibers With Large Diffusers
Brief Title: Surgery and Photodynamic Therapy in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Todd Demmy, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269674; RPCI-RP-9812
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; recurrent malignant mesothelioma; epithelial mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Chemotherapy, Adjuvant; Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adjuvant therapy — Lung surgery
Procedure: conventional surgery — Lung surgery
Drug: porfimer sodium — iv

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill cancer cells. Combining photodynamic therapy with surgery may be an effective treatment for malignant mesothelioma.

PURPOSE: Phase II trial to study the effectiveness of combining photodynamic therapy with surgery in treating patients who have malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of adjuvant photodynamic therapy with large diffuser fibers in patients with malignant mesothelioma undergoing surgery.
* Compare results of this regimen in these patients to historical controls.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a pilot study.

Patients receive porfimer sodium IV over 5-10 minutes on day 1. Patients undergo pleurectomy or pleuropneumonectomy followed by intracavitary photodynamic therapy on day 3.

Patients are followed at 1 month, every 4 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant mesothelioma, including the following cell types:

  * Mixed mesothelial
  * Sarcomatous
* Stage I or II disease using the Butchart system as determined by CT scan or MRI
* Disease confined to 1 hemithorax
* No tumor involvement of esophagus or heart as evidenced by CT scan

  * Pericardial or diaphragmatic involvement allowed if disease is limited to the ipsilateral chest
  * N2 disease allowed if no contralateral pleural involvement
* No adenocarcinoma or nonmesothelioma sarcoma of the chest wall

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.5 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 3.0 mg/dL
* Alkaline phosphatase less than 2 times upper limit of normal (ULN)
* SGOT less than 2 times ULN

Renal

* Creatinine less than 3.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months

Pulmonary

* Arterial partial pressure of carbon dioxide (pCO_2) less than 50 torr at rest
* Predicted postoperative FEV_1 at least 800 mL with maximum oxygen consumption/kg at least 15 mL/min
* Predicted postoperative total lung capacity at least 40% of hemoglobin and alveolar ventilation

Other

* Not pregnant
* No other concurrent malignancy except nonmelanoma skin cancer
* No contraindication to general anesthetic
* No history of porphyria
* No indicated sensitivity to porfimer sodium

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 30 days since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest
* No prior radiotherapy for mesothelioma

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1999-03; Primary Completion 2006-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 month, every 4 months for 2 years, and then every 6 months for 3 years
Comparison of results from this regimen to historical controls | At completion of study
Toxic effects | 1 month, every 4 months for 2 years, and then every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Todd L. Demmy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States